CLINICAL TRIAL: NCT07310589
Title: A Randomized Controlled Trial to Evaluate the Effects of a Visual-Interactive LINE Chatbot on Self-Management of EGFR-TKI-Related Side Effects in Patients With Lung Cancer
Brief Title: Effects of a Visual Interactive LINE Chatbot on Self-Management of EGFR-TKI Related Side Effects in Patients With Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202506172RINB
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: LINE Chatbot; EGFR-TKIs; side effects; Self-management ability; Quality of life; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either an intervention group receiving usual care plus access to a visual interactive LINE chatbot or a control group receiving usual care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LINE Chatbot Intervention Group (Experimental): Participants receive usual care plus access to a visual interactive LINE chatbot designed to support self-management of treatment-related side effects during EGFR-TKI therapy.
  Interventions: Behavioral: Visual-Interactive LINE Chatbot
- usual care (No Intervention): Participants receive usual care, which consists of standard paper-based educational materials provided as part of routine clinical care, without access to the LINE chatbot.

INTERVENTIONS:
Behavioral: Visual-Interactive LINE Chatbot — Participants receive access to a visual-interactive LINE chatbot designed to support self-management of EGFR-TKI-related side effects. The chatbot provides interactive and visualized educational content, symptom monitoring guidance, and self-care recommendations throughout the treatment period, in addition to usual care.
  Arms: LINE Chatbot Intervention Group

SUMMARY:
This study aims to evaluate a visual interactive LINE chatbot designed to support self-management of treatment-related side effects among patients with advanced lung cancer receiving epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) therapy.

Patients receiving EGFR-TKI treatment often experience long-term side effects that require ongoing self-management. In this randomized controlled trial, participants will be assigned to receive either usual care alone or usual care plus access to the LINE chatbot intervention, which provides visualized and interactive educational content for symptom monitoring and self-care.

The primary outcome of this study is self-management ability related to EGFR-TKI-associated side effects. Secondary outcomes include quality of life during treatment and overall satisfaction with the LINE chatbot intervention.

DETAILED DESCRIPTION:
The objective of this study is to evaluate a visual interactive LINE chatbot designed to support self-management of treatment-related side effects among patients with advanced lung cancer receiving epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) therapy.

This study uses a randomized controlled trial design. Participants will be recruited from a medical center in northern Taiwan and randomly assigned to either an intervention group or a control group. The control group will receive standard education and routine clinical care, while the intervention group will receive standard care plus access to the visual interactive LINE chatbot intervention. The chatbot provides visualized and interactive educational content to support symptom monitoring and self-care during treatment.

Assessments will be conducted at baseline and at multiple follow-up time points after enrollment to evaluate self-management ability related to EGFR-TKI-associated side effects, quality of life during treatment, and overall satisfaction with the chatbot intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage IIIB to IVB unresectable or inoperable non-small cell lung cancer (NSCLC), or those with first disease recurrence who are receiving oral targeted therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, with the ability to perform self-care activities.
* Patients receiving epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) therapy, including gefitinib, erlotinib, afatinib, dacomitinib, or osimertinib.
* Willingness to participate in the study, with completion of the informed consent process and provision of written informed consent.
* Ability to communicate in Chinese and to independently operate a smartphone and use the LINE application.

Exclusion Criteria:

* Patients diagnosed with a second primary malignancy or multiple malignancies.
* Patients receiving other anticancer treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-Management Ability（PAM-13） | at baseline and at 1, 3, and 6 months post-intervention
  Self-management ability is measured using the Patient Activation Measure (PAM-13) developed by Hibbard et al. (2005).
  The PAM-13 consists of 13 items assessing an individual's knowledge, skills, and confidence in managing their health or chronic condition.
  Each item is rated on a 4-point Likert scale, and raw scores are transformed into a standardized score ranging from 0 to 100, with higher scores indicating greater self-management ability and willingness to engage in self-care.
  The Chinese version of the PAM-13 has demonstrated good internal consistency, with a Cronbach's alpha of 0.835.

SECONDARY OUTCOMES:
Quality of Life Related to EGFR-TKI Treatment（FACT-EGFRI-18） | at baseline and at 1, 3, and 6 months post-intervention
  Quality of life is assessed using the Functional Assessment of Cancer Therapy-Epidermal Growth Factor Receptor Inhibitor 18-item scale (FACT-EGFRI-18) developed by Wagner et al. (2013).
  The FACT-EGFRI-18 consists of 18 items evaluating the impact of EGFR-TKI-related dermatologic toxicities on patients' physical, psychological, social, skin, nail, and hair-related well-being.
  Items are rated on a 5-point Likert scale, with total scores ranging from 18 to 90.
  Higher scores indicate greater symptom burden and poorer quality of life. The Chinese version of the FACT-EGFRI-18 has demonstrated good internal consistency, with Cronbach's alpha values ranging from 0.83 to 0.95.
Overall User Satisfaction With the LINE Chatbot Intervention (CSQ-8) | At 3 months after the intervention
  User satisfaction is measured using the Client Satisfaction Questionnaire-8 (CSQ-8) developed by Larsen et al. (1979).
  The CSQ-8 consists of 8 items assessing overall satisfaction with healthcare or psychosocial interventions.
  Each item is rated on a 4-point Likert scale, with total scores ranging from 8 to 32, where higher scores indicate greater satisfaction with the intervention.
  The CSQ-8 has demonstrated high internal consistency, with reported Cronbach's alpha values ranging from 0.93 to 0.95.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographic characteristics, intervention assignment, and outcome measure scores (self-management ability, quality of life, and user satisfaction), will be shared. A data dictionary and related study documentation will also be made available. Data will be shared upon reasonable request after publication of the primary study results.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after publication of the primary study results and will be available for a period of five years.
Access Criteria: Researchers who provide a methodologically sound research proposal may request access to the data. Requests will be reviewed by the study investigators, and access will be granted following approval and execution of a data use agreement.

REFERENCES:
- [Result] Lim SM, Shiau CWC, Cheng LJ, Lau Y. Chatbot-Delivered Psychotherapy for Adults With Depressive and Anxiety Symptoms: A Systematic Review and Meta-Regression. Behav Ther. 2022 Mar;53(2):334-347. doi: 10.1016/j.beth.2021.09.007. Epub 2021 Oct 12. PMID 35227408
- [Result] Plachouri KM, Florou V, Georgiou V, Georgiou S. Cutaneous Side Effects of Modern Targeted Therapy and Immunotherapy in Patients with Dermatological Malignancies. Cancers (Basel). 2023 Jun 9;15(12):3126. doi: 10.3390/cancers15123126. PMID 37370736
- [Result] Galmarini E, Marciano L, Schulz PJ. The effectiveness of visual-based interventions on health literacy in health care: a systematic review and meta-analysis. BMC Health Serv Res. 2024 Jun 11;24(1):718. doi: 10.1186/s12913-024-11138-1. PMID 38862966
- [Result] Dan H, Jiang Q, Jia X, Qi G, Zong D, Li Z. Dermatologic toxicities in epidermal growth factor receptor: a comprehensive pharmacovigilance study from 2013 to 2023. Front Med (Lausanne). 2024 Jan 24;10:1283807. doi: 10.3389/fmed.2023.1283807. eCollection 2023. PMID 38327269